CLINICAL TRIAL: NCT04859114
Title: Effect of Presenting Survival Information as Text or Pictograph During Periviable Birth
Brief Title: Effect of Presenting Survival Information as Text or Pictograph During Periviable Birth Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Mir A Basir, Associate Professor of Pediatrics, Medical College of Wisconsin
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 2021-121
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Premature Birth
Keywords: decision making; neonatal resuscitation; risk communication; prenatal counseling
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: 2x3 between subjects
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Text-only outcome data, 30% survival (Active Comparator): Participants in this arm are provided a repeat of the outcome data in a text-only format, displaying a 30% chance of survival.
  Interventions: Behavioral: Format of outcome data presentation; Behavioral: Displayed chance of survival
- Text-only outcome data, 60% survival (Active Comparator): Participants in this arm view a repeat of the outcome data in a text-only format, displaying a 60% chance of survival.
  Interventions: Behavioral: Format of outcome data presentation; Behavioral: Displayed chance of survival
- Static pictograph outcome data, 30% survival (Experimental): Participants in this arm view a static pictograph displaying the outcome data and showing a 30% chance of survival.
  Interventions: Behavioral: Format of outcome data presentation; Behavioral: Displayed chance of survival
- Static pictograph outcome data, 60% survival (Experimental): Participants in this arm view a static pictograph displaying the outcome data and showing a 60% chance of survival.
  Interventions: Behavioral: Format of outcome data presentation; Behavioral: Displayed chance of survival
- Iterative pictograph outcome data, 30% survival (Experimental): Participants in this arm view an iterative pictograph displaying the outcome data and showing a 30% chance of survival.
  Interventions: Behavioral: Format of outcome data presentation; Behavioral: Displayed chance of survival
- Iterative pictograph outcome data, 60% survival (Experimental): Participants in this arm view an iterative pictograph displaying the outcome data and showing a 60% chance of survival.
  Interventions: Behavioral: Format of outcome data presentation; Behavioral: Displayed chance of survival

INTERVENTIONS:
Behavioral: Format of outcome data presentation — Outcome data is provided to participants as either text-only, a static pictograph, or an iterative pictograph.
Behavioral: Displayed chance of survival — In the outcome data provided to participants, they view either a 30% or 60% chance of survival.

SUMMARY:
Women recruited from the internet will be put in a hypothetical situation of being in labor at 22 weeks of pregnancy, and presented with information on the likelihood of survival and chance of disability for babies born at this gestational age.

Participants will be randomized to receive this outcome data in one of three formats: as text-only, in a static pictograph, or in an iterative pictograph. Participants will also be randomized to seeing the chance of survival as 30% or 60%.

Participants were then asked to choose between comfort care and intensive care in this situation. Participants' religiosity, value of the sanctity of life, and health literacy were also assessed.

DETAILED DESCRIPTION:
A recent study by Kidszun et al. (2020) concluded that for mothers placed in a hypothetical situation of choosing between comfort care and intensive care at 22 weeks gestation, treatment choice was not influenced by the chance of survival. Specifically, there was no difference in treatment choice between moms who were told the baby would have a 30% chance of survival and moms who were told the baby would have a 60% chance of survival.

The study was conducted using a written vignette that included a paragraph on the chance of survival and the chance of disability among the survivors.

In this study, we will adapt the vignette the Kidszun et al. (2020) team used, and provide it to an internet-based sample of women. In this vignette, participants will be put in a hypothetical situation of being in labor at 22 weeks of pregnancy, provided a description of the treatment choices of intensive care or comfort care, and provided data on outcome information at this gestational age.

After reading the vignette, participants will be randomized to view either: a repeat of the text information on outcome data, a static pictograph, or an iterative pictograph. Participants will also be randomized to seeing the chance of survival as 30% or 60%, making this a 2 (chance of survival) x 3 (data presentation format) between-subjects experiment.

After viewing a repeat of the outcome information, participants will be asked to choose between intensive care or comfort care for their hypothetical child. We will also collect information on values, religiosity, health literacy, subjective numeracy, a subjective probability estimate, and demographics.

ELIGIBILITY:
Inclusion Criteria:

Women who have:

* had a child,
* are currently of child-bearing age (defined as 18-45)
* and who live in the U.S.

Exclusion Criteria:

* Minors
* Those unable to read English
* Those who only could complete the survey on their phone. (For formatting purposes, a tablet or computer is necessary.)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The survey was distributed only to women.
Enrollment: 1052 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonnell SM, Basir MA, Yan K, Liegl MN, Windschitl PD. Effect of Presenting Survival Information as Text or Pictograph During Periviable Birth Counseling: A Randomized, Controlled Trial. J Pediatr. 2023 Jun;257:113382. doi: 10.1016/j.jpeds.2023.02.026. Epub 2023 Mar 7. PMID 36894129

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text-only Outcome Data, 30% Survival | Text-only Outcome Data, 60% Survival | Static Pictograph Outcome Data, 30% Survival | Static Pictograph Outcome Data, 60% Survival | Iterative Pictograph Outcome Data, 30% Survival | Iterative Pictograph Outcome Data, 60% Survival
Started | 176 | 177 | 179 | 177 | 176 | 167
Completed | 176 | 177 | 179 | 177 | 176 | 167
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Text-only Outcome Data, 30% Chance of Survival: Participants in this arm are provided a 30% chance of survival seen by repeat of the outcome data in a text-only format.
  Displayed chance of survival: In the outcome data provided to participants, they view either a 30% or 60% chance of survival.
  Format of outcome data presentation: Outcome data is provided to participants as either text-only, a static pictograph, or an iterative pictograph.
- Static Pictograph Outcome Data, 30% Chance of Survival: Participants in this arm are provided a 30% chance of survival seen by a static pictograph displaying the outcome data.
  Displayed chance of survival: In the outcome data provided to participants, they view either a 30% or 60% chance of survival.
  Format of outcome data presentation: Outcome data is provided to participants as either text-only, a static pictograph, or an iterative pictograph.
- Iterative Pictograph Outcome Data, 30% Survival: Participants in this arm are provided a 30% chance of survival, seen by an iterative pictograph displaying the outcome data.
  Displayed chance of survival: In the outcome data provided to participants, they view either a 30% or 60% chance of survival.
  Format of outcome data presentation: Outcome data is provided to participants as either text-only, a static pictograph, or an iterative pictograph.
- Text-only Outcome Data, 60% Chance of Survival: Participants in this arm are provided a 60% chance of survival seen by repeat of the outcome data in a text-only format.
  Displayed chance of survival: In the outcome data provided to participants, they view either a 30% or 60% chance of survival.
  Format of outcome data presentation: Outcome data is provided to participants as either text-only, a static pictograph, or an iterative pictograph.
- Static Pictograph Outcome Data, 60% Chance of Survival: Participants in this arm are provided a 60% chance of survival seen by a static pictograph displaying the outcome data.
  Displayed chance of survival: In the outcome data provided to participants, they view either a 30% or 60% chance of survival.
  Format of outcome data presentation: Outcome data is provided to participants as either text-only, a static pictograph, or an iterative pictograph.
- Iterative Pictograph Outcome Data, 60% Survival: Participants in this arm are provided a 60% chance of survival, seen by an iterative pictograph displaying the outcome data.
  Displayed chance of survival: In the outcome data provided to participants, they view either a 30% or 60% chance of survival.
  Format of outcome data presentation: Outcome data is provided to participants as either text-only, a static pictograph, or an iterative pictograph.
- Total: Total of all reporting groups
Arm/Group | Text-only Outcome Data, 30% Chance of Survival | Static Pictograph Outcome Data, 30% Chance of Survival | Iterative Pictograph Outcome Data, 30% Survival | Text-only Outcome Data, 60% Chance of Survival | Static Pictograph Outcome Data, 60% Chance of Survival | Iterative Pictograph Outcome Data, 60% Survival | Total
Number analyzed (Participants) | 176 | 179 | 176 | 177 | 177 | 167 | 1052
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (7.9) | 34.1 (7.0) | 34.1 (7.2) | 34.6 (8.0) | 33.8 (7.7) | 33.6 (7.4) | 34.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 179 | 176 | 177 | 177 | 167 | 1052
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 26 | 32 | 28 | 27 | 24 | 172
  Not Hispanic or Latino | 136 | 148 | 140 | 144 | 140 | 136 | 844
  Unknown or Not Reported | 5 | 5 | 4 | 5 | 10 | 7 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 3 | 2 | 4 | 2 | 16
  Asian | 7 | 16 | 8 | 8 | 13 | 8 | 60
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 1 | 0 | 3
  Black or African American | 27 | 25 | 32 | 33 | 20 | 32 | 169
  White | 132 | 133 | 127 | 129 | 135 | 120 | 776
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 5 | 5 | 4 | 5 | 28
Region of Enrollment [Number; unit: participants]
  United States | 176 | 179 | 176 | 177 | 177 | 167 | 1052
Education [Count of Participants; unit: Participants]
  8th grade or less | 1 | 2 | 4 | 0 | 0 | 2 | 9
  9th-12th grade, no diploma | 14 | 5 | 8 | 11 | 9 | 5 | 52
  High school diploma or equivalent | 44 | 46 | 39 | 33 | 39 | 45 | 246
  Some college | 16 | 20 | 23 | 25 | 26 | 20 | 130
  2-year college degree | 10 | 22 | 15 | 13 | 14 | 20 | 94
  4-year college degree | 47 | 52 | 54 | 57 | 41 | 45 | 296
  Graduate or professional degree | 44 | 31 | 33 | 37 | 47 | 27 | 219
  Preferred not to answer | 0 | 1 | 0 | 1 | 1 | 3 | 6
Previous Neonatal Intensive Care Unit exposure [Count of Participants; unit: Participants]
  Yes | 43 | 47 | 51 | 58 | 51 | 46 | 296
  No | 127 | 129 | 122 | 103 | 117 | 114 | 712
  Do not know | 4 | 3 | 3 | 10 | 7 | 4 | 31
  Prefers not to answer | 2 | 0 | 0 | 6 | 2 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Hypothetical Treatment Choice
Description: Participant's hypothetical treatment choice of either palliative care or intensive care. Participants are told: "If the child was actually born shortly after the conversation described above, which treatment would you prefer if you were in this situation?" and given the options of "Palliative care treatment" or "Intensive care treatment". This variable is assessed for the frequency of each option chosen.
Time Frame: Assessed immediately post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Text-only Outcome Data, 30% Survival | Text-only Outcome Data, 60% Survival | Static Pictograph Outcome Data, 30% Survival | Static Pictograph Outcome Data, 60% Survival | Iterative Pictograph Outcome Data, 30% Survival | Iterative Pictograph Outcome Data, 60% Survival
Number analyzed (Participants) | 176 | 177 | 179 | 177 | 176 | 167
Participants
  Chose intensive care | 130 | 135 | 143 | 126 | 129 | 123
  Chose palliative care | 46 | 42 | 36 | 51 | 47 | 44

2. Secondary Outcome: Values: Quality of Life or Sanctity of Life
Description: Participants answered the following: "In making end-of-life decisions: 1) Quality of life is much more important than preserving life, 2) Quality of life is somewhat more important than preserving life, 3) Preserving life is somewhat more important than quality of life, or 4) Preserving life is much more important than quality of life." In the range of 1-4, a score of 4 indicated the greatest participant value of sanctity of life.
Time Frame: Assessed post-intervention, immediately after treatment choice.
Measure: Count of Participants; unit: Participants
Arm/Group | Text-only Outcome Data, 30% Survival | Text-only Outcome Data, 60% Survival | Static Pictograph Outcome Data, 30% Survival | Static Pictograph Outcome Data, 60% Survival | Iterative Pictograph Outcome Data, 30% Survival | Iterative Pictograph Outcome Data, 60% Survival
Number analyzed (Participants) | 176 | 177 | 179 | 177 | 176 | 167
Participants
  Quality of life is much more important | 80 | 90 | 85 | 93 | 90 | 78
  Quality of life is somewhat more important | 42 | 45 | 42 | 47 | 38 | 44
  Preserving life is somewhat more important | 31 | 26 | 30 | 21 | 31 | 26
  Preserving life is much more important | 23 | 16 | 22 | 16 | 17 | 19

3. Secondary Outcome: Preference for Medical Autonomy
Description: Participants were asked on a 4-point scale their medical autonomy preferences, in the form of: "In making medical decisions... 1) I always prefer to have the doctor make medical decisions for me. 2) I would prefer to have the doctor make medical decisions for me most of the time. 3) I would prefer to make my own medical decisions most of the time. 4) I always prefer to make my own decisions."
Time Frame: Assessed post-intervention, immediately after treatment choice
Measure: Count of Participants; unit: Participants
Arm/Group | Text-only Outcome Data, 30% Survival | Text-only Outcome Data, 60% Survival | Static Pictograph Outcome Data, 30% Survival | Static Pictograph Outcome Data, 60% Survival | Iterative Pictograph Outcome Data, 30% Survival | Iterative Pictograph Outcome Data, 60% Survival
Number analyzed (Participants) | 176 | 177 | 179 | 177 | 176 | 167
Participants
  Responded "I always prefer to have the doctor make medical decisions for me." | 36 | 49 | 46 | 42 | 53 | 48
  Responded "I would prefer to have the doctor make medical decisions for me most of the time." | 43 | 55 | 44 | 58 | 44 | 35
  Responded "I would prefer to make my own medical decisions most of the time." | 64 | 41 | 53 | 49 | 46 | 60
  Responded "I always prefer to make my own decisions." | 33 | 32 | 36 | 28 | 33 | 24

4. Secondary Outcome: Subjective Sense of Probability
Description: After reporting an objective value of the probability of survival that has been described to them in the vignette and intervention, participants report their subjective sense of probability.
  Specifically, they will read: "Assume again that your baby was born prematurely at 22 weeks and given intensive care treatment. The doctor gave you the same information you read earlier. At a gut level, what would you believe is your own baby's actual chance of survival? Please click somewhere along the bar below to indicate your response." Participants use a slider scale below the item to respond from "No chance of survival" to "Definitely will survive". Responses will be coded numerically on a 100-point scale, with 0 representing "No chance of survival" to 100 representing "Definitely will survive".
Time Frame: Assessed post-intervention, immediately after treatment choice.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Text-only Outcome Data, 30% Survival | Text-only Outcome Data, 60% Survival | Static Pictograph Outcome Data, 30% Survival | Static Pictograph Outcome Data, 60% Survival | Iterative Pictograph Outcome Data, 30% Survival | Iterative Pictograph Outcome Data, 60% Survival
Number analyzed (Participants) | 176 | 177 | 179 | 177 | 176 | 167
units on a scale | 61.5 (29.9) | 66.1 (25.0) | 64.8 (27.7) | 65.4 (25.9) | 65.7 (26.7) | 62.7 (26.0)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Description: This was a minimal risk study, with randomization to hypothetical information for a questionnaire based study, i.e. not a biological intervention. All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Text-only Outcome Data, 30% Survival | Text-only Outcome Data, 60% Survival | Static Pictograph Outcome Data, 30% Survival | Static Pictograph Outcome Data, 60% Survival | Iterative Pictograph Outcome Data, 30% Survival | Iterative Pictograph Outcome Data, 60% Survival
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT04859114/Prot_SAP_000.pdf